CLINICAL TRIAL: NCT03008525
Title: Vitamin D and Its Metabolites Quantification in Adipose Tissues of Obese and Non-obese
Brief Title: Vitamin D and Its Metabolites Quantification in Adipose Tissues of Obese and Non-obese Patients.
Acronym: VITADOSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-23
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Endocrine
MeSH Terms: conditions — Obesity | interventions — Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obese patients (group OB) (Experimental): patients with body mass index ≥ 35 kg/m²
  Interventions: Biological: subcutaneous and visceral adipose tissue biopsies; Biological: blood samples analysis
- non-obese patients (group NO) (Active Comparator): patients with body mass index < 30 kg/m²
  Interventions: Biological: subcutaneous and visceral adipose tissue biopsies; Biological: blood samples analysis

INTERVENTIONS:
Biological: subcutaneous and visceral adipose tissue biopsies — Subcutaneous and visceral adipose tissue biopsies during operation
Biological: blood samples analysis — Blood sampling is required to measure plasma cholecalciferol, calcidiol and calcitriol concentrations, as well as biological parameters of interest.
  Another plasma/serum tube is used to measure pro- and anti-inflammatory cytokines and adiponectin.

SUMMARY:
Vitamin D (VD) is a pleiotropic hormone, involved in many physiological processes including calcium and phosphorus absorption. The VD metabolism begin to be well-known and involves a hepatic hydroxylation (mediated by enzymes, which belong to the cytochrome P450 family) leading to the production of the 25(OH)D, which corresponds to the circulating form of the VD. After circulation in blood, the 25(OH)D is submitted to a second hydroxylation in the kidney resulting to the generation of 1,25(OH)2D, the active metabolite of VD. Numerous epidemiological studies reported an inverse relationship between obesity and circulation level of 25(OH)D. Several mechanisms could explain the low level of 25(OH)D observed in obese subjects, the more classical evoked being based on sequestration and/or dilution of VD in adipose tissue (AT), the main VD storage site. However, this mechanism has never been demonstrated. In order to confirm this hypothesis, the concentration of VD and its metabolites in adipose tissue need to be quantified.

The objective of this study is to determine the concentration of VD and its metabolites in adipose tissue as well as adipose tissue mass quantification and distribution (visceral or subcutaneous) to highlight putative difference of VD and its metabolites quantities between obese and non-obese patients. A quantification of VD metabolism, inflammation and lipid metabolism gene expression will be realized on biopsies. Correlations between gene expression and quantity of VD in tissue will be carrying out.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a BMI greater than 35 kg / m2 (group OB) or less than 30 kg / m² (group NO)
* Subject undergoing bariatric surgery (OB group) or abdominal surgery (group NO)

Exclusion Criteria:

* Regular intake of dietary supplements or vitamin supplements in the last three months
* For the subjects of the group NO:

  * Malnourished patient (BMI <18.5 kg / m2, weight loss greater than 5% in 1 month or 10% in 6 months)
  * Subject with an infection or inflammatory syndrome (CRP> 10 mg / L and / or white blood cells> 12000 / mm3)
  * Non-cancerous subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2025-09-13 (Estimated); Study Completion 2026-09-13 (Estimated)

PRIMARY OUTCOMES:
quantification of VD and its metabolites on subcutaneous and visceral adipose tissue biopsies | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France